CLINICAL TRIAL: NCT03146390
Title: Essential Oils With and Without Alcohol: in Vivo Antibacterial Effect
Brief Title: Essential Oils With and Without Alcohol: Substantivity and Antiplaque Effect
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Inmaculada Tomas, Senior Lecturer, University of Santiago de Compostela
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 023/2017
Record Dates: First submitted 2017-04-30; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Oral Biofilm; Dental Plaque; Periodontitis
Keywords: biofilms; essential oils; microscopy, confocal; mouthwashes
MeSH Terms: conditions — Dental Plaque; Periodontitis | interventions — Oils, Volatile; Ethanol; Water

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Essential oils (Listerine Mentol) (Active Comparator): 1. a single mouthwash with 20 ml of essential oils for 30 seconds
  2. 20 ml rinses for 30 seconds with essential oils/2 times daily (1/0/1).
  Interventions: Drug: Essential oils
- Water (Placebo Comparator): 1. a single mouthwash with 20 ml of sterile water for 30 seconds
  2. 20 ml rinses for 30 seconds with sterile water/2 times daily (1/0/1).
  Interventions: Other: Water
- Alcohol free essential oils (Experimental): 1. a single mouthwash with 20 ml of alcohol free essential oils for 30 seconds
  2. 20 ml rinses for 30 seconds with alcohol free essential oils/2 times daily (1/0/1).
  Interventions: Drug: Alcohol free essential oils

INTERVENTIONS:
Drug: Essential oils — all subjects will perform all interventions of all arms
  Other Names: Listerine Mentol
  Arms: Essential oils (Listerine Mentol)
Drug: Alcohol free essential oils — all subjects will perform all interventions of all arms
  Other Names: Listerine Zero
  Arms: Alcohol free essential oils
Other: Water — all subjects will perform all interventions of all arms
  Other Names: Sterile Water
  Arms: Water

SUMMARY:
The Essential oils (EO) are composed by a wide diversity of products. Therefore, their antimicrobial activity will be related to their composition, configuration, amount and their possible interaction. The traditional formulation containing EO (T-EO) is a complex mixture of phenolic compounds combined with determinate EO: 0.092% of eucalyptol, 0.064% of thymol, 0.06% of methyl-salicylate and y 0.042% of menthol. All of this solved in a hydroalcoholic vehicle containing from a 21.6% to a 26.9% of alcohol. Thus, T-EO contain ethanol, which is a chemical compound used in order to dissolve and stabilize the numerous substances present in the rinse. The concentration of ethanol present in the T-EO rinses, as previously said, is more than 20%. This concentration of ethanol, higher than 20%, is been found sufficient to dissolve the EO but insufficient to have a direct antibacterial effect. In fact, the manufacturer presents the alcohol contain (21.6%), among others, as an inactive ingredient in its formula. Over the years, the adequacy of the use of ethanol in mouthwashes, as well as their effects on the surfaces of composite restorations and their possible role in development of oropharyngeal cancer have been discussed. Although a direct cause-and-effect correlation between the development of oropharyngeal carcinoma and the use of alcohol-based rinses has not been demonstrated and probably it will never be (at least by epidemiological studies), it is considered desirable to eliminate ethanol from daily mouthwashes, especially for those patients at higher risk. Furthermore, the fact that the alcohol is present in its formula, have produced that some clinical practitioners do not prescribe the traditional formula due to the controversy of the issue. All this have lead to the development of new, alcohol free formulations of EO (Af-EO).

The composition of the Af-EO is exactly the same in their active ingredients (Eucalyptol, Thymol, Methyl-salycilate and Menthol), but sodium fluoride has been added. Some differences are found in their inactive ingredients. These are based on the alcohol containing of the T-EO, without presence in the Af-EO and the presence of Propylene Glycol, sodium lauryl sulfate and sucralose in the Af-EO, without presence in the T-EO.

In order to measure the efficacy of a mouthwash against the dental plaque two different concepts should be defined: the substantivity and antiplaque effect. The substantivity of an oral antiseptic is defined as the prolonged adherence to the oral surfaces and its slow release at effective doses which guarantee the persistence of the antimicrobial activity. The more substantivity an oral antiseptic has the better. For its study in vivo, the most popular models are those which analyze the effect that a single mouthwash has in a mature biofilm.

The second aspect that should be studied from an oral antiseptic, the antiplaque effect, is defined as the capacity that an agent has to avoid the formation of bacterial aggregates (plaque) on the oral surfaces. For its study in vivo, models start from a baseline sample with levels of plaque near to 0 in order to assess the power of the antiseptic to reduce the formation of bacterial plaque (normally dental plaque) against the control. A clinical study of 6 months using a determinate antiplaque agent is necessary in order to tag an antiseptic as effective. However, in the literature, there is an established model of 4 days of plaque regrowing which can assess the inhibitory activity that the mouthwashes have per se; furthermore, it determines the relative efficacy of the different formulations being considered as predictable of the antiplaque effect of an antiseptic.

In addition, another important factor in the study in vivo of an oral antiseptic is the necessity to conserve intact the oral biofilm at all stages: formation, recollection and analysis of the oral samples. This is in order not to interfere the delicate three dimensional structure of the oral biofilm which has been proven to be essential in the resistance to the effects of an external antiseptic agent. For these reasons, the study of the oral biofilm with the help of intraoral disks hold in specially designed apparatus combined with the application of the Confocal Laser Scanning Microscopy have proved to be very valuable at the study of the oral biofilm in its intact hydrated natural state.

Since an alcohol free formulation of the EO have come up to the market, it seems convenient to compare its effects to the traditional one. Although some studies comparing the effects of T-EO and Af-EO have been found, none of them assessed and compared their substantivity and antiplaque effect in an in vivo model of structured oral biofilm. For this reason, the aim of the present study was to compare the in vivo antibacterial effect (immediate effect, substantivity and antiplaque effect) of the EO with and without alcohol in structured oral biofilm.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy adults.
* Minimum of 24 permanent teeth.
* No gingivitis (Community Periodontal Index score = 0).
* No periodontitis (Community Periodontal Index score = 0).
* Absence of untreated caries.

Exclusion Criteria:

* Smoker or former smoker.
* Presence of dental prostheses.
* Presence of orthodontic devices.
* Antibiotic treatment or routine use of oral antiseptics in the previous 3 months.
* Presence of any systemic disease that could alter the production or composition of saliva.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-07-31 (Estimated); Study Completion 2017-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Bacterial viability (%) (substantivity) | Baseline, 30 seconds, 1 hour, 3 hours, 5 hours and 7 hours after the single application
  ratio of alive/dead bacteria
Bacterial viability (%) (antiplaque effect) | 10 hours after the last mouthwash
  ratio of alive/dead bacteria
Change in the Biofilm Thickness (Microns) (substantivity) | baseline, 30 seconds, 1 hour, 3 hours, 5 hours and 7 hours after the single application
  thickness of the biofilm from the base of the substrate to the top surface of the biofilm
Biofilm Thickness (Microns) (Antiplaque effect) | 10 hours after the last mouthwash
  thickness of the biofilm from the base of the substrate to the top surface of the biofilm
Covering Grade (%) (antiplaque effect) | 10 hours after the last mouthwash
  area of the substrate that is covered by the biofilm after the 4 days of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Quintas V, Prada-Lopez I, Donos N, Suarez-Quintanilla D, Tomas I. Antiplaque effect of essential oils and 0.2% chlorhexidine on an in situ model of oral biofilm growth: a randomised clinical trial. PLoS One. 2015 Feb 17;10(2):e0117177. doi: 10.1371/journal.pone.0117177. eCollection 2015. PMID 25689859
- [Background] Quintas V, Prada-Lopez I, Prados-Frutos JC, Tomas I. In situ antimicrobial activity on oral biofilm: essential oils vs. 0.2 % chlorhexidine. Clin Oral Investig. 2015 Jan;19(1):97-107. doi: 10.1007/s00784-014-1224-3. Epub 2014 Apr 1. PMID 24687247